CLINICAL TRIAL: NCT07060456
Title: A Phase III, Multicenter, Randomized, Double Blinded, Parallel-controlled Study Comparing the Efficacy and Safety of HRS9531 Versus Placebo in Subjects With Type 2 Diabetes Mellitus Inadequately Controlled With Basal Insulin.
Brief Title: Efficacy and Safety of HRS9531 in Participants With Type 2 Diabetes Treated With Basal Insulin
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fujian Shengdi Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HRS9531-305
Record Dates: First submitted 2025-06-22; First posted 2025-07-11 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-04

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment group A: HRS9531-low dose (Experimental)
  Interventions: Drug: HRS9531
- Treatment group B: HRS9531-high dose (Experimental)
  Interventions: Drug: HRS9531
- Treatment group C (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HRS9531 — HRS9531-low dose
  Arms: Treatment group A: HRS9531-low dose
Drug: HRS9531 — HRS9531-high dose
  Arms: Treatment group B: HRS9531-high dose
Drug: Placebo — Placebo
  Arms: Treatment group C

SUMMARY:
The study is being conducted to evaluate the efficacy and safety of HRS9531 compared with placebo in participants with type 2 diabetes mellitus not adequately controlled with basal insulin, with or without metformin and/or sodium-glucose cotransporter-2 (SGLT2) inhibitor. The study may include up to 23 visits.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, able and willing to provide a written informed consent
2. Diagnosed with type 2 diabetes ≥ 90 days；
3. On stable once-daily dose of basal insulin alone or in combination with metformin and/or SGLT2 inhibitor ≥ 90 days;
4. HbA1c was 7.5%~11.0% (both inclusive);
5. Body Mass Index (BMI) ≥22 kg/m2 at screening.

Exclusion Criteria:

1. A history of type 1 diabetes, specific diabetes, or secondary diabetes;
2. Have a history of severe hypoglycemia within t180 days prior to screening;
3. History of acute cardiovascular and cerebrovascular diseases within 180 days prior to screening；
4. Have a history of malignancy within 5 years;
5. Known or suspected allergy or intolerance to the investigational medicinal products or related products;
6. Participation in any clinical trial of an approved or non-approved investigational product/treatment within the last 90 days;
7. Any conditions that the Investigator judges might not be suitable to participate in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-07-25 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Change in HbA1c | from baseline to Week 40
  Change in HbA1c after 40 weeks of treatment.

SECONDARY OUTCOMES:
Proportion of subjects reaching HbA1<7.0% | from baseline to Week 40
  Proportion of subjects reaching HbA1<7.0% after 40 weeks of treatment.
Proportion of subjects reaching HbA1≤6.5% | from baseline to Week 40
  Proportion of subjects reaching HbA1≤6.5% after 40 weeks of treatment.
Change in FPG | from baseline to Week 40
  Change in FPG after 40 weeks of treatment.
Change in Diabetes Treatment Satisfaction Questionnaire (DTSQ) Score | From baseline to Week 40
  Change from baseline in DTSQs after 40 weeks of treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Perking University Peoples' Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided